CLINICAL TRIAL: NCT06364956
Title: A Phase Ib/II Prospective Study to Evaluate the Safety and Efficacy of the Combination of Neoadjuvant Palbociclib and Tislelizumab in Platinum-refractory cT2-4aN0M0 Bladder Urothelial Carcinoma.
Brief Title: Clinical Trail of Neoadjuvant of Tislelizumab Combined With Palbociclib in Patients With Platinum-refractory Bladder Urothelial Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-124-02
Record Dates: First submitted 2024-03-06; First posted 2024-04-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer
Keywords: Tislelizumab; Palbociclib; neoadjuvant; bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase Ib clinical trial (Experimental): Tislelizumab, 200mg q3W, combined with two predefined dose groups of palbociclib: 100mg QD and 125mg QD, separately.
  Interventions: Drug: Tislelizumab combined with two predefined dose groups of palbociclib
- Phase II clinical trial (Experimental): Tislelizumab, 200mg q3W, combined with RP2D dose of palbociclib was selected for phase II clinical trial.
  Interventions: Drug: RP2D dose Of Tislelizumab combined with palbociclib was selected for phase II clinical trial.

INTERVENTIONS:
Drug: Tislelizumab combined with two predefined dose groups of palbociclib — Tislelizumab, 200mg q3W, combined with two predefined dose groups of palbociclib: 100mg QD and 125mg QD, separately.
  Arms: Phase Ib clinical trial
Drug: RP2D dose Of Tislelizumab combined with palbociclib was selected for phase II clinical trial. — After the exploration of Tislelizumab, 200mg q3W combined with palbociclib, and the maximal tolerated dose (MTD) was determined, then RP2D dose of Tislelizumab combined with palbociclib was selected for phase II clinical trial.
  Arms: Phase II clinical trial

SUMMARY:
In order to explore the safety and antitumor efficacy of different doses of CDK4/6 inhibitor Palbociclib in combination with the Tislelizumab in platinum-refractory cT2-4aN0M0 bladder urothelial carcinoma, a phase Ib/II study was conducted.

This study will adopt a 3+3 design and include two predefined dose groups of palbociclib: 100mg QD, 125mg QD. Initially, Tislelizumab, 200 mg administered by intravenous infusion on Day 1 of each 21-day will be administered in combination. The trial will use the first cycle (28 days) as the observation period for tolerability, observing and evaluating the occurrence of DLTs after medication and determining the maximum tolerated dose/maximum administered dose (MTD/MAD) and recommended phase 2 dose (RP2D) of the combination therapy (30 patients) .

This study provide further evidence for improving the efficacy of neoadjuvant treatment forplatinum-refractory cT2-4aN0M0 bladder urothelial carcinoma and to offer new options for precision treatment of bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in this study, able to provide written informed consent and can understand and agree to comply with the requirements of the study and schedule of assessments.
2. Aged over 18 years on day of signing informed consent
3. Patients with urothelial bladder cancer, having residual lesions following TURBT surgery, staged cT2-T4aN0M0 as histologically confirmed and radiologically assessed based on the TNM Staging System for Bladder Cancer of American Joint Committee on Cancers (AJCC) ; predominantly histological classification of urothelial carcinoma (at least 50%) for patients with mixed-histology bladder cancer.
4. Patients with mutations or copy number variation (CNV) alterations, such as CDKN2A, CDKN2B CNV deletion, indicating the activation of cell cycle-related pathways.
5. ECOG Performance Status 0 or 1
6. Ineligible for Cisplatin treatment as judged by investigator. Patients who are ineligible for Cisplatin chemotherapy should meet at least one of the following criteria: ECOG performance status > 1 or Karnofsky performance status 60% to 70%; creatinine clearance less than 60 mL/min; ≥ Grade 2 hearing loss according to NCI-CTCAE v5.0; ≥ Grade 2 neuropathy peripheral according to NCI-CTCAE v5.0; ≥ Grade 3 cardiac failure according to New York Heart Association Cardiac Function Classification
7. Patients will receive radical cystectomy following neoadjuvant therapy as assessed by investigator, meet surgical indication and are willing to receive the surgery.
8. Tumor tissue samples collected during TURBT must be available, and relevant pathological reports are required. Fresh surgical tissue samples or pathological slides are optional
9. Have adequate organ function as indicated by the following screening laboratory values (obtained ≤ 14 days prior to enrollment):

   a.Patients must not be administered with growth factors ≤ 14 days prior to sampling for the screening tests of: i.Absolute neutrophil count ≥ 1.5 x 109/L ii.Platelets ≥ 90 x 109/L iii.Hemoglobin ≥ 90 g/L b.International normalized ratio or activated partial thromboplastin time ≤ 1.5 x upper limit of normal (ULN).

   c.Serum total bilirubin ≤ 1.5 x ULN (≤ 3 x ULN, if Gilbert's syndrome or if indirect bilirubin concentrations were suggestive of extrahepatic source of the elevation).

   e.Aspartate transaminase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 2.5 x ULN f.Patients can tolerate major abdominal surgery as suggested by pulmonary function test results
10. Unpregnant females or females of childbearing potential must be willing to use a highly effective contraceptive method for the duration of the study, and ≥ 120 days after the last dose of Tislelizumab or chemotherapy agents, whichever is later, and have a negative urine or serum pregnancy test ≤ 7 days prior to enrollment.

Exclusion Criteria:

1. Received prior therapies targeting PD-1, PD-L1, PD-L2, CTLA4, or other antibodies or drugs specifically targeting T-cell costimulation or checkpoint pathways.
2. Received other approved systemic anticancer therapies or systemic immunomodulators (including but not limited to interferon, interleukin 2, and tumor necrosis factor) within 28 days prior to enrollment.
3. Received prior radiotherapy for bladder cancer.
4. Received anticancer drug therapies with the following exceptions:

   1. For patients who have received prior systemic chemotherapy, a treatment-free interval of at least 12 months from the last dose of chemotherapy until the start of neoadjuvant therapy is required
   2. Local intravesical chemotherapy or immunotherapy must be discontinued at least 1 week before start of the investigational neoadjuvant medication treatment
5. Received major surgery or had major trauma within 28 days prior to enrollment (vascular access placement and TURBT are not considered as major surgeries).
6. Severe chronic or active infections requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to enrollment (HBV infection will be ruled out according to Exclusion Criteria # 12).
7. Received live vaccines within 28 days prior to enrollment (seasonal vaccines for influenza are generally inactivated vaccines and are allowed. Intranasal vaccines are live vaccines and are not allowed.)
8. Active autoimmune diseases that requires systemic treatment and may impact study treatment as assessed by investigator
9. Any condition that requires extensive chronic treatment with either hormones or any other immunosuppressive medications that may impact study treatment as assessed by investigator.
10. With history of potassium, sodium, calcium abnormalities or hypoalbuminemia, interstitial lung disease, pneumonitis or history of uncontrolled systemic diseases, including diabetes, hypertension, cardiovascular diseases (such as active cardiac diseases within 6 months prior to enrollment, including: severe/unstable angina pectoris, myocardial infarction, symptomatic congestive heart failure, and ventricular arrhythmia requiring medical treatment) that may impact study treatment as assessed by investigator.
11. HBV Patients with untreated chronic hepatitis B or hepatitis B virus (HBV) carriers with HBV DNA ≥ 500 IU/mL (2500 copies/mL) cannot be enrolled. Note: inactive hepatitis B surface antigen (HBsAg) carriers and patients who received continuous antiviral treatments and have stable active hepatitis B infection (HBV DNA < 500 IU/mL or < 2500 copies/mL) can be enrolled. HBV DNA testing will be performed only for patients testing positive for antibody to hepatitis B core antigen (anti-HBc).
12. Patients with active hepatitis C cannot be enrolled. Patients with a negative HCV antibody test at Screening or positive HCV antibody test followed by a negative HCV RNA test at Screening can be enrolled. The HCV RNA test will be performed only for patients testing positive for HCV antibody.
13. History of immunodeficiency (including human immunodeficiency virus [HIV] positive, other acquired, congenital immunodeficiency diseases) or history of allogeneic stem cell transplantation or organ transplantation.
14. Known hypersensitivity to other monoclonal antibodies.
15. Known hypersensitivity to any investigational agents or their excipients.
16. Patients with toxicities or AEs (as a result of any prior treatment) which have not recovered to baseline or stabilized, except for toxicities or AEs not considered a likely safety risk (eg, alopecia, neuropathy, and specific laboratory abnormalities) as assessed by investigator.
17. Underlying medical conditions or alcohol or drug abuse or dependence that were to be unfavorable for the administration of investigational agents or may have affected the interpretation of the results or rendered the patient at high risk from treatment complications.
18. Concurrent participation in another therapeutic clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Phase I: The safety dose of the combination of Tislelizumab and Palbociclib | 12 months
  The study aims to evaluate the safety dose of the combination of Tislelizumab combined with palbociclib in patients with cT2-4aN0M0 bladder cancer. The safety dose was according to "3+3" dose escalation principle.
  Participants with dose-limiting toxicity (DLT) as assessed by NCI CTC 5.0 and the administered drug dose.
Phase II: Percentage of Participants With Pathological Complete Response(pCR) | 24 months
  Pathological evaluation of the resected tumor tissue and regional lymph nodes showed no residual tumor cells, complete disappearance of the tumor lesions, and no evidence of new lesions.

SECONDARY OUTCOMES:
Percentage of Participants With Pathological Downstaging(pDS) | 24 months
  The pathological downstaging rate is defined as the evaluation of whether the staging is degraded to ≤ T2 based on the post-surgery pathological findings. The rates of cT2N0 → pT0N0, cT3-4aN0 → pT0N0, cT2N0 → ≤ pT1N0, cT3-4aN0 → ≤ pT1N0 will be calculated, and the 2 sided Clopper-Pearson 95% confidence interval (CI) of pathological downstaging rate will be calculated to assess the precision of the estimated pathological downstaging rate.
Event-free survival (EFS) | 24 months
  Event-free survival (EFS) was determined from start date of the first dose of neoadjuvant treatment to date of disease progression, death from any cause, or onset of other tumors.
overall survival (OS) | 24 months
  OS was measured from the date the participant started study to death for any reason.
Safety and AE | 24 months
  Number of unique patients who had a treatment-related (possible, probable, or definite) adverse event using the Medical Dictionary for Regulatory Activities (MedDRA) terms and graded per NCI-CTCAE v5.0.
  Number and Grade of patients who had a surgery-related adverse event (surgery-related AE) will be measured according to the Clavien-Dindo classification.

OTHER OUTCOMES:
Biomarker Endpoint Analyses | 24 months
  To explore biomarkers in urine, blood, and tumor tissues (collected from TURBT) at baseline and tissue samples collected from radical cystectomy. Biomarkers include PD-L1, Ki67 expression in tumor tissues, immune cells profiling and gene expression and tumor mutation profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Tianxin Lin, Ph.D, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (8):
- China (8):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan